CLINICAL TRIAL: NCT03567733
Title: Prospective Registry of Patients Over 75 Years Old Treated With Xience Sierra Stents". Sierra 75 Study
Brief Title: Prospective Registry of Patients Over 75 Years Old Treated With Xience Sierra Stents. Sierra 75 Study
Acronym: SIERRA 75
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: SIERRA 75 EPIC-05
Record Dates: First submitted 2018-06-12; First posted 2018-06-26 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease
Keywords: Dual antiplatelet treatment; Elderly patients
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease: Drug- eluting Stent
  Interventions: Device: XIENCE Sierra

INTERVENTIONS:
Device: XIENCE Sierra — Percutaneous coronary intervention

SUMMARY:
This prospective registry is intended to evaluate the safety and efficacy of the XIENCE Sierra stent.

DETAILED DESCRIPTION:
This prospective registry is intended to analyze clinical outcomes in elderly patients treated with XIENCE Sierra stent and in pre-established subgroups (stable and unstable coronary artery disease).

ELIGIBILITY:
Inclusion Criteria:

* Age> 75 years.
* With indication of percutaneous revascularization.
* Presence of de novo coronary artery lesions located in a native coronary artery.
* Informed consent signed

Exclusion Criteria:

* Cardiogenic shock at the time of the PCI(Percutaneous Coronary Intervention)
* Cardiac arrest before the PCI
* Life expectancy of the patient under 1 year
* Participation in another study with a drug or device in clinical research
* Clinical decision that excludes the use of drug-eluting stents
* Confirmed allergy to aspirin and / or thienopyridines.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients older than 75 years with de novo native coronary artery lesions, candidate to undergo revascularisation with a coronary device.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Safety.The composite of cardiac death, myocardial infarction (MI) and stent thrombosis (Academic Research Consortium definitive/probable). . | 12 month
  The composite of cardiac death, myocardial infarction (MI) and stent thrombosis (Academic Research Consortium definitive/probable).
  .
Efficacy.The incidence of clinically driven target lesion revascularization (TLR). | 12 month
  The incidence of clinically driven target lesion revascularization (TLR).

SECONDARY OUTCOMES:
All death. | 12 month
  All death.
  Systemic embolism, Major bleeding event (BARC ≥ 2)
Cardiac death. | 12 month
  Cardiac death.
Target Vessel revascularization. | 12 month
  Target Vessel revascularization.
Target lesion revascularization. | 12 month
  Target lesion revascularization.
Stent thrombosis (ARC definite/probable). | 12 month
  Stent thrombosis (ARC definite/probable).
Major bleeding event (BARC type 2-5). | 12 month
  Major bleeding event (BARC type 2-5).
Stroke. | 12 month
  Stroke.
Procedural success. | 12 month
  Procedural success ( Residual stenosis <30% after implantation at the narrowest point of the treated vascular segment).
Rate of patients with DAPT. | 1 month
  Rate of patients with DAPT.
Rate of patients with DAPT. | From 1 to 3 months
  Rate of patients with DAPT.
Rate of patients with DAPT. | From 3 to 6 months
  Rate of patients with DAPT.
Rate of patients with DAPT. | From 6 to 12 months
  Rate of patients with DAPT.
Collection of imaging data by Optical coherence tomography (OCT). | 12 month
  Collection of imaging data by OCT.
Collection of imaging data by Intravascular Ultrasound (IVUS). | 12 month
  Collection of imaging data by IVUS.

CONTACTS AND LOCATIONS:
Locations (44):
- Portugal (7):
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar Lisboa Occidental. Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE, Espinho
  - Hospital do Espírito Santo de Évora, Evora
  - Hospital Do Divino Espirito Santo De Ponta Delgada, Ponta Delgada
  - Hospital Do Divino Espirito Santo, Ponta Delgada
  - Centro Hospitalar de Setubal, EPE - Hospital Sao Bernardo, Setúbal
- Spain (37):
  - Hospital Universitario Vinalopo, Elche, Alicante
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital de Mérida, Mérida, Badajoz
  - Hospital Universitari Germans Trias I Pujol de Badalona, Badalona, Barcelona
  - Hospital de Puerto Real, Puerto Real, Cádiz
  - Hospital Universitari Son Espases, Palma de Mallorca, Mallorca
  - Hospital General Universitario de Albacete, Albacete
  - Hospital Universitario San Juan de Alicante, Alicante
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Puerta Del Mar, Cadiz
  - Hospital Galdakao-Usansolo, Galdakao
  - Hospital de Cabueñes, Gijón
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complejo Hospitalario Regional de Málaga, Málaga
  - Hospital Clinico Universitario Virgen de La Arrixaca, Murcia
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen de La Salud, Toledo
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari I Politècnic La Fe, Valencia
  - Hospital Universitario Álvaro Cunqueiro, Vigo
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa F, van Klaveren D, James S, Heg D, Raber L, Feres F, Pilgrim T, Hong MK, Kim HS, Colombo A, Steg PG, Zanchin T, Palmerini T, Wallentin L, Bhatt DL, Stone GW, Windecker S, Steyerberg EW, Valgimigli M; PRECISE-DAPT Study Investigators. Derivation and validation of the predicting bleeding complications in patients undergoing stent implantation and subsequent dual antiplatelet therapy (PRECISE-DAPT) score: a pooled analysis of individual-patient datasets from clinical trials. Lancet. 2017 Mar 11;389(10073):1025-1034. doi: 10.1016/S0140-6736(17)30397-5. PMID 28290994
- [Background] Valgimigli M, et al. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2017 Aug 26
- [Background] Kedhi E, Stone GW, Kereiakes DJ, Serruys PW, Parise H, Fahy M, Simonton CA, Sudhir K, Sood P, Smits PC. Stent thrombosis: insights on outcomes, predictors and impact of dual antiplatelet therapy interruption from the SPIRIT II, SPIRIT III, SPIRIT IV and COMPARE trials. EuroIntervention. 2012 Sep;8(5):599-606. doi: 10.4244/EIJV8I5A92. PMID 22995087
- [Background] de Belder A, de la Torre Hernandez JM, Lopez-Palop R, O'Kane P, Hernandez Hernandez F, Strange J, Gimeno F, Cotton J, Diaz Fernandez JF, Carrillo Saez P, Thomas M, Pinar E, Curzen N, Baz JA, Cooter N, Lozano I, Skipper N, Robinson D, Hildick-Smith D; XIMA Investigators. A prospective randomized trial of everolimus-eluting stents versus bare-metal stents in octogenarians: the XIMA Trial (Xience or Vision Stents for the Management of Angina in the Elderly). J Am Coll Cardiol. 2014 Apr 15;63(14):1371-5. doi: 10.1016/j.jacc.2013.10.053. Epub 2013 Nov 21. PMID 24216285
- [Background] Gao L, Hu X, Liu YQ, Xue Q, Wang Y. Comparison of coronary DES and BMS in octogenarians: A systematic review and meta-analysis. J Geriatr Cardiol. 2013 Dec;10(4):336-43. doi: 10.3969/j.issn.1671-5411.2013.04.004. PMID 24454326
- [Background] Urban P, Meredith IT, Abizaid A, Pocock SJ, Carrie D, Naber C, Lipiecki J, Richardt G, Iniguez A, Brunel P, Valdes-Chavarri M, Garot P, Talwar S, Berland J, Abdellaoui M, Eberli F, Oldroyd K, Zambahari R, Gregson J, Greene S, Stoll HP, Morice MC; LEADERS FREE Investigators. Polymer-free Drug-Coated Coronary Stents in Patients at High Bleeding Risk. N Engl J Med. 2015 Nov 19;373(21):2038-47. doi: 10.1056/NEJMoa1503943. Epub 2015 Oct 14. PMID 26466021
- [Background] Morice MC, Talwar S, Gaemperli O, Richardt G, Eberli F, Meredith I, Zaman A, Fajadet J, Copt S, Greene S, Urban P. Drug-coated versus bare-metal stents for elderly patients: A predefined sub-study of the LEADERS FREE trial. Int J Cardiol. 2017 Sep 15;243:110-115. doi: 10.1016/j.ijcard.2017.04.079. Epub 2017 Apr 25. PMID 28579168
- [Result] de la Torre Hernandez JM, Palop RL, Jimenez Mazuecos JM, Saez PC, Gutierez-Barrios A, Pinar E, Cid B, Fernandez L, Camarero TG, Urbano-Carrillo C, Oteo Dominguez JF, Jimenez Diaz VA, Gomez Menchero AE, Fernandez EG, Cordoba Soriano JG, Ocaranza R, Ucar EA, Roman KGS, Leal S, Caceres GM, Linares Vicente JA, Ferre GF, Carrillo X, Rama Merchan JC, Costa C, Sanchis J, Fernandes R, Rodrigues A, Vegas Valle JM, Pereira H, de Prado AP. Prospective application of a bleeding and ischemic risks-adjusted antithrombotic protocol in elderly patients revascularized with everolimus-eluting stents: EPIC05-Sierra75 study. J Geriatr Cardiol. 2022 May 28;19(5):354-366. doi: 10.11909/j.issn.1671-5411.2022.05.009. PMID 35722037
- See also: Related Info — http://www.precisedaptscore.com/predapt/webcalculator.html
- See also: Study Results — https://doi.org/10.11909/j.issn.1671-5411.2022.05.009